CLINICAL TRIAL: NCT03101904
Title: The Effect of Chronic Nitrate Supplementation on Acute Mountain Sickness and Exercise Performance in Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangor University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: Jan 27 2016
Record Dates: First submitted 2016-03-10; First posted 2017-04-05 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrate then Placebo (Experimental): Participants will consume a daily a beetroot shot for six days. Each shot will consist of: 1x70ml concentrated NO-3 shot of rich Beetroot juice (~7mmol nitrate; Beet It, James White Drinks Ltd, Ipswich, UK).
  Following a minimum of ten days wash out, participants will then consume a daily Nitrate-depleted beetroot shot for six days. Each shot will consist of 1x70ml nitrate-depleted beetroot Placebo shot (~0.003mmol of nitrate; Beet It, James White Drinks Ltd, Ipswich, UK).
  Interventions: Dietary Supplement: Beetroot Juice; Dietary Supplement: Placebo
- Placebo then Nitrate (Placebo Comparator): Participants will consume a daily Nitrate-depleted beetroot shot for six days. Each shot will consist of 1x70ml nitrate-depleted beetroot Placebo shot (~0.003mmol of nitrate; Beet It, James White Drinks Ltd, Ipswich, UK).
  Following a minimum of ten days wash out, participants will then consume a daily beetroot shot for six days. Each shot will consist of: 1x70ml concentrated NO-3 shot of rich Beetroot juice (~7mmol nitrate; Beet It, James White Drinks Ltd, Ipswich, UK).
  Interventions: Dietary Supplement: Beetroot Juice; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beetroot Juice
  Other Names: Nitrate-rich beetroot juice
Dietary Supplement: Placebo
  Other Names: Nitrate-depleted beetroot juice

SUMMARY:
The study will aim to describe and evaluate the effect of chronic beetroot juice supplementation on acute mountain sickness symptoms and exercise in a hypoxic environment. It is hypothesized that beetroot supplementation will decrease acute mountain sickness and increase exercise performance.

ELIGIBILITY:
Inclusion Criteria:

* Women only: Regular menstrual cycle or post-menopausal

Exclusion Criteria:

* Stayed at altitude above 2500m in the last 6 months
* Traveled to altitude above 2500m in the last 2 months
* Unable to give informed consent
* Unstable medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-02; Primary Completion 2017-01-09 (Actual); Study Completion 2017-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie H Macdonald, PhD, Principal Investigator — Bangor University
Locations (1):
- School of Sport, Health and Exercise Sciences, Bangor University, Bangor, Gwynedd, United Kingdom

REFERENCES:
- [Result] Sampson JB, Kobrick JL, Johnson RF. Measurement of subjective reactions to extreme environments: the Environmental Symptoms Questionnaire. Military Psychology. 1994; 6(4):215-233. doi: 10.1207/s15327876mp0604_2

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1. Participants completed a baseline demographics visit including the following assessments:
     * Age
     * Height
     * Body mass
     * Blood pressure
     * Haemoglobin
     * Normoxic VO2max (maximal exercise) test
  2. Participants then completed a minimum 48 h wash out
  3. Participants completed a hypoxic VO2max test at 14.1% O2
Groups:
- Nitrate First, Then Placebo: Participants will consume a daily a beetroot shot for six days. Each shot will consist of: 1x70ml concentrated NO-3 shot of rich Beetroot juice (~7mmol nitrate; Beet It, James White Drinks Ltd, Ipswich, UK).
  10 day wash out.
  Following a minimum of ten days wash out, participants will then consume a daily Nitrate-depleted beetroot shot for six days. Each shot will consist of 1x70ml nitrate-depleted beetroot Placebo shot (~0.003mmol of nitrate; Beet It, James White Drinks Ltd, Ipswich, UK).
- Placebo First, Then Nitrate: Participants will consume a daily Nitrate-depleted beetroot shot for six days. Each shot will consist of 1x70ml nitrate-depleted beetroot Placebo shot (~0.003mmol of nitrate; Beet It, James White Drinks Ltd, Ipswich, UK).
  10 day wash out.
  Following a minimum of ten days wash out, participants will then consume a daily beetroot shot for six days. Each shot will consist of: 1x70ml concentrated NO-3 shot of rich Beetroot juice (~7mmol nitrate; Beet It, James White Drinks Ltd, Ipswich, UK).
Period: First Intervention (6 Days)
Arm/Group | Nitrate First, Then Placebo | Placebo First, Then Nitrate
Started | 13 | 10
Baseline Bloods (Day 1) | 13 | 10
AMS Trial (Day 5) | 13 | 10
Performance Trial (Day 6) | 13 | 10
Completed | 13 | 10
Not Completed | 0 | 0
Period: Wash Out (10 Days)
Arm/Group | Nitrate First, Then Placebo | Placebo First, Then Nitrate
Started | 13 | 10
Completed | 10 | 10
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Period: Second Intervention (6 Days)
Arm/Group | Nitrate First, Then Placebo | Placebo First, Then Nitrate
Started | 10 | 10
Baseline Bloods (Day 1) | 10 | 10
AMS Trial (Day 5) | 10 | 10
Performance Trial (Day 6) | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population is different from overall number because it does not include the 3 participants that did not complete the study.
Groups:
- Nitrate First, Then Placebo: Participants consumed a daily a beetroot shot for six days. Each shot will consist of: 1x70ml concentrated NO-3 shot of rich Beetroot juice (~7mmol nitrate; Beet It, James White Drinks Ltd, Ipswich, UK).
  10 day wash out
  After a minimum 10-day wash-out, participants consumed a daily Nitrate-depleted beetroot shot for six days. Each shot will consist of 1x70ml nitrate-depleted beetroot Placebo shot (~0.003mmol of nitrate; Beet It, James White Drinks Ltd, Ipswich, UK).
- Placebo First, Then Nitrate: Participants consumed a daily Nitrate-depleted beetroot shot for six days. Each shot will consist of 1x70ml nitrate-depleted beetroot Placebo shot (~0.003mmol of nitrate; Beet It, James White Drinks Ltd, Ipswich, UK).
  10 day wash out
  After a minimum 10-day wash-out, participants consumed a daily a beetroot shot for six days. Each shot will consist of: 1x70ml concentrated NO-3 shot of rich Beetroot juice (~7mmol nitrate; Beet It, James White Drinks Ltd, Ipswich, UK).
- Total: Total of all reporting groups
Arm/Group | Nitrate First, Then Placebo | Placebo First, Then Nitrate | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (4) | 22 (4) | 22 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 10 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Maximal Aerobic Capacity [Mean (Standard Deviation); unit: ml/kg/min] | 53 (6) | 50 (6) | 51 (6)

OUTCOME MEASURES:

1. Primary Outcome: Acute Mountain Sickness (AMS-C) as Assessed by the Environmental Symptoms Questionnaire.
Description: Acute Cerebral Mountain Sickness score (AMS-C) calculated from the 11-item Environmental Symptoms Questionnaire (ESQ; Sampson et al., 1994). Participants rate the severity of each item from zero to five, and the ratings were multiplied by their factorial loadings and summed.
  Unabbreviated scale title: Acute Cerebral Mountain Sickness Abbreviated title: AMS-C Unit of measure: Scores on a scale Minimum value: 0 Maximum value: 5 Interpretation: Higher scores mean a worse outcome
Time Frame: Measured on the fifth day of supplementation with a six-hour exposure to hypoxia
Measure: Mean (Standard Error); unit: scores on a scale
Groups:
- Nitrate: Participants consumed a daily a beetroot shot for six days. Each shot will consist of: 1x70ml concentrated NO-3 shot of rich Beetroot juice (~7mmol nitrate; Beet It, James White Drinks Ltd, Ipswich, UK).
- Placebo: Participants consumed a daily Nitrate-depleted beetroot shot for six days. Each shot will consist of 1x70ml nitrate-depleted beetroot Placebo shot (~0.003mmol of nitrate; Beet It, James White Drinks Ltd, Ipswich, UK).
Arm/Group | Nitrate | Placebo
Number analyzed (Participants) | 20 | 20
scores on a scale | 0.36 (0.09) | 0.21 (0.04)

2. Secondary Outcome: Hypoxic Exercise Performance as Assessed by Time to Exhaustion at 80% of Hypoxic V̇O2max Reserve.
Description: On day six of each supplementation protocol, participants completed a time to exhaustion test at 80% of their hypoxic V̇O2max reserve in acute hypoxia (FiO2 14.1%, equivalent 3225 m). Maximal exercise performance is defined as time to exhaustion (TTE) determined by the time from onset of test to task failure (volitional exhaustion or inability to maintain treadmill speed).
Time Frame: Measured on the sixth day of supplementation
Population: Five participants did not complete the TTE on day 6 because of injury or technical reasons, e.g., cramp or tripping while on the treadmill, and one of these was also removed from analyses relating to RPE on day 5 because of failure to use the RPE scale consistently.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Nitrate | Placebo
Number analyzed (Participants) | 15 | 15
seconds | 666 (206) | 656 (184)

ADVERSE EVENTS:
Time Frame: Adverse even data was collected throughout participant involvement in the study. Adverse even data was collected 2 hours and 48 hours after each laboratory visit.
Arm/Group | Nitrate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/20
Other Adverse Events (participants affected / at risk) | 1/23 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitrate (N=23) | Placebo (N=20)
Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Possible inter-costal muscle strain or pericarditis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-10-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT03101904/SAP_000.pdf
  • Informed Consent Form (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/04/NCT03101904/ICF_001.pdf